CLINICAL TRIAL: NCT00559221
Title: Fludarabine and Cytarabine as Continuous Infusion Plus Idarubicin With Granulocyte-Colony Stimulating Factor (G-CSF) Priming for Patients Younger Than 60 Years With Resistant Acute Myeloid Leukemia
Brief Title: FLAG+Ida With G-CSF Priming for Patients Younger Than 60 Years With Resistant AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-007A
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2007-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Ida-FLAG protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention)
  Interventions: Drug: FLAG+IDA

INTERVENTIONS:
Drug: FLAG+IDA — Fludarabine, cytarabine, G-CSF

SUMMARY:
- To determine the feasibility of fludarabine and cytarabine as continuous infusion plus idarubicin with granulocyte-colony stimulating factor priming for patients with resistant acute myeloid leukemia other than acute promyelocytic leukemia

DETAILED DESCRIPTION:
- The feasibility will be evaluated in terms of toxicities, complete remission rate, duration of complete remission, disease-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Failure to achieve CR after initial induction chemotherapy including standard dose cytarabine.
* Early relapse, occurring after a first CR lasting less than 12 months.
* Patients with multiple relapses will be included.
* Written informed consent must be given.
* 15 and 60 years of age.
* 2 or less by ECOG performance scale.

Exclusion Criteria:

* acute promyelocytic leukemia
* pregnant or lactating

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2004-12; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate, duration of complete remission, toxicities | 06/2008

SECONDARY OUTCOMES:
progression-free survival, overall survival | 06/2008

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, professor, Principal Investigator — Ulsan Universtity Hospital, ROK
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Lee JH, Joo YD, Bae SH, Lee JH, Kim DY, Lee WS, Ryoo HM, Jo JC, Choi Y, Lee KH; CoOperative Study Group A for Hematology (COSAH). A prospective, multicenter phase II study of continuous infusion of FLAG for patients older than 60 yr with resistant acute myeloid leukemia: a comparison with intensive younger patients' trial. Eur J Haematol. 2016 Feb;96(2):188-97. doi: 10.1111/ejh.12568. Epub 2015 May 6. PMID 25891993